CLINICAL TRIAL: NCT07127185
Title: Individualized Precision Therapy With Ceftobiprole Guided by PK/PD in Geriatric Populations
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Wu Jionghui, Dr., Chinese PLA General Hospital
Other Study IDs: S2025-448-01
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Ceftobiprole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ceftobiprole: Clinical Blood Sampling Protocol for Ceftobiprole in Geriatric Patients: Elderly patients received intravenous ceftobiprole (250 mg or 500 mg) every 12 hours, with infusion durations of 1 h, 1.5 h, or 2 h. After 3 days of antibiotic therapy (steady-state achievement), blood sampling was performed as follows:
  Trough Concentration: A 3-mL peripheral blood sample was collected from the antecubital vein pre-dose (before the next scheduled administration) using EDTA-containing Vacutainers®.
  Peak Concentration: A blood sample was drawn immediately after completion of the intravenous infusion. All blood specimens were centrifuged at 2500 × g for 10 minutes. Plasma samples were stored at -20°C and analyzed within 1 week of collection via liquid chromatography-tandem mass spectrometry (LC-MS/MS).
  Interventions: Diagnostic Test: LS/MS

INTERVENTIONS:
Diagnostic Test: LS/MS — Quantitative determination of ceftobiprole concentrations in plasma and urine was performed using liquid chromatography-tandem mass spectrometry (LC-MS/MS).

SUMMARY:
Ceftobiprole, a fifth-generation cephalosporin, exhibits potent antibacterial activity against MRSA, penicillin-resistant Streptococcus pneumoniae (PRSP), and certain Gram-negative bacteria (e.g., Pseudomonas aeruginosa). In elderly patients, significant interindividual variability often leads to inappropriate dosing (subtherapeutic or excessive), compromising efficacy or increasing toxicity risks. This prospective, multicenter study will enroll patients aged ≥60 years receiving ceftobiprole. Using LC-MS/MS for therapeutic drug monitoring (TDM), we will measure plasma concentrations and integrate individual characteristics (age, body weight, creatinine clearance, etc.). Population pharmacokinetic (PPK) modeling with Bayesian forecasting will be employed to estimate individual PK parameters and identify covariates influencing variability, thereby establishing a PPK model for ceftobiprole in the elderly.

Based on pathogen-specific MIC values, dosing regimens (dose, frequency) will be dynamically optimized to guide precision therapy. Subsequent TDM data will continuously refine the PPK model, creating a self-optimizing system. This framework lays the groundwork for extending individualized treatment strategies to other antimicrobials in geriatric populations.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥60 years Scheduled to receive ceftobiprole therapy for >5 days No prior ceftobiprole use within 1 month before enrollment

Exclusion Criteria:

* Patients requiring renal replacement therapy (hemodialysis, peritoneal dialysis, or continuous renal replacement therapy [CRRT]) or with renal impairment history (nephrectomy, renal transplantation, solitary kidney, uremia) Obese patients with body mass index (BMI) ≥30 kg/m²

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Professional Translation for Clinical Research Protocols: Enroll patients aged ≥60 years receiving ceftobiprole therapy at Chinese PLA General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-12 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Ceftobiprole Concentration | after 3 days of antibiotic therapy
  Plasma Ceftobiprole Concentration and Urinary Ceftobiprole Concentration

IPD SHARING:
Plan to Share IPD: No
Unauthorized disclosure of the research protocol may undermine investigator motivation and compromise scientific validity.